CLINICAL TRIAL: NCT04575155
Title: Development & Pilot of the Technology-Enabled Alliance for Medication Therapy Management
Acronym: TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Gordon and Betty Moore Foundation (Other); Walgreens (Industry); ACCESS Community Health Network (Other)
Responsible Party: Principal Investigator, Michael S. Wolf, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 8036
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Polypharmacy
Keywords: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAM Strategy (Experimental): Patients randomized to the TEAM intervention arm will receive at least one call from a Walgreens pharmacist to help them with their complex Rx regimens. Pharmacists will have read/write EHR access with established Epic security points. Through shared access to patients' medical records, pharmacists can perform comprehensive medication therapy management services, document and communicate patients' Rx challenges for review and action by primary care providers. After the pharmacist calls the patient for a Comprehensive Medication Review, they will add notes in their medication list for the prescriber, requesting the removal or discontinuation of prescribed drugs that patients report they are not taking and adding medications omitted from the provider's list. The pharmacist will provide notifications via secured Epic messaging direct to prescribers of any patient concerns.The prescriber will make changes to the patient's EHR and/or contact the patient as they see fit.
  Interventions: Behavioral: TEAM Strategy
- Enhanced Usual Care (No Intervention): Patients randomized to enhanced usual care will have the medical record available to a Walgreens pharmacist with 'read only' access. All patients at the five targeted health centers already have read-only access in place. This means the Walgreens pharmacist will have the capability to review a patient's record as necessary. The pharmacist may refer to the EHR as needed and in a reactive manner; such as if a patient were to request a medication requiring review for billing purposes (i.e. verify insurance, prior authorizations), or if a patient safety concern was raised (e.g. potential drug-drug or drug- disease interaction, therapeutic duplication, etc.). Similarly, read only EHR access means pharmacists must continue to use existing communication channels (e.g. phone, fax) to contact prescribers.

INTERVENTIONS:
Behavioral: TEAM Strategy — 1. Pharmacists will have read/write EHR access with established Epic security points
  2. Pharmacists will initiate medication reconciliation activities by calling the patient for a Comprehensive Medication Review. Pharmacists will add notes in their medication list for the prescriber, requesting the removal or discontinuation of prescribed drugs that patients report they are not taking and adding medications omitted from the provider's list. The pharmacist will provide notifications via secured Epic messaging direct to prescribers of any patient concerns.
  3. At 6 month if poor adherence is determined, the pharmacist will initiate Therapy Management Review which is a call from the pharmacist to the patient specifically about the medication(s) for which they have poor adherence. If necessary, the pharmacist will create notes and send an in-basket message to the prescriber.
  4. The prescriber will make changes to the patient's EHR and/or contact the patient as they see fit.
  Arms: TEAM Strategy

SUMMARY:
The investigators will link community pharmacy and primary care practices via a shared electronic health record to improve medication therapy management for older patients taking complex prescription (Rx) regimens. The Technology-Enabled Alliance for Medication Therapy Management (TEAM) intervention will link a major, national community pharmacy chain (Walgreens) to primary care practices (Access Community Health Network) via a shared electronic health record (EHR) platform (Epic, Verona WI). Through shared access to patients' medical records, pharmacists can perform comprehensive medication therapy management services, document and communicate patients' Rx challenges for review and action by primary care providers. The aims of this investigation are to:

1. Evaluate the fidelity and efficacy of the TEAM intervention to promote healthcare provider counseling, medication reconciliation, and safe regimen use among adults taking complex Rx regimens.
2. Explore patient, healthcare provider (pharmacist, prescriber), community pharmacy and/or primary care practice barriers to implementation.
3. Determine the costs of the TEAM intervention from both a community pharmacy and primary care practice perspective.

DETAILED DESCRIPTION:
The investigators will link community pharmacy and primary care practices via a shared electronic health record to improve medication therapy management for older patients taking complex prescription (Rx) regimens. The Technology-Enabled Alliance for Medication Therapy Management (TEAM) intervention will link a major, national community pharmacy chain (Walgreens) to primary care practices (ACCESS community health network) via a shared electronic health record (EHR) platform (Epic, Verona WI). Through shared access to patients' medical records, pharmacists can perform comprehensive medication therapy management services, document and communicate patients' Rx challenges for review and action by primary care providers.

The investigators will conduct a 2-arm pilot to evaluate the efficacy of the TEAM intervention compared to enhanced usual care. The investigators will enroll a total of 120 English and Spanish-speaking patients prescribed five or more chronic medications. Enrolled patients will complete a follow-up interview two months after their baseline interview.

The TEAM intervention enables a pharmacist to help patients on complex Rx regimens via medication reviews by telephone and clinical decision support. Pharmacists will call patients to conduct a Comprehensive Medication Review (CMR). Pharmacists will be able to document and communicate patients' medication challenges for review and action by primary care providers. A CMR will:

1. Ensure the primary care physician knows all medications the patient is taking (reconciliation)
2. Investigate if patients are taking medication as prescribed, in a safe manner (proper use)
3. Monitor and detect any drug-related adverse effects (ADEs) (surveillance)
4. Address any questions or concerns patients may have about their medicine (e.g. side effects, treatment alternatives, dietary restrictions, cost, 90 vs. 30 day scripts; education)
5. Inquire about patients' adherence to regimens, what barriers they may experience (e.g. cost, forgetfulness) and if they need assistance (e.g. synchronization requests, pill box or reminder tools, etc.; adherence).

After performing the CMR, the pharmacist will provide timely notifications via secure, EHR-based messaging direct to prescribers of any medication concerns, based on either 1) pharmacy information (e.g. medications ordered by other prescribers, fill data), 2) patient report of problems during phone-based encounters, or 3) pharmacist review of the patient record.

The aims of this investigation are to:

1. Evaluate the fidelity and efficacy of the TEAM intervention to promote healthcare provider counseling, medication reconciliation, and safe regimen use among adults taking complex Rx regimens.
2. Explore patient, healthcare provider (pharmacist, prescriber), community pharmacy and/or primary care practice barriers to implementation.
3. Determine the costs of the TEAM intervention from both a community pharmacy and primary care practice perspective.

ELIGIBILITY:
1. Patient is age 50 and older
2. Patient is English or Spanish speaking
3. Patient has established care at one of the involved ACCESS health centers (defined as 1 visit within 18 months)
4. Patient is an existing Walgreens customer (had 1 or more medications filled at collocated Walgreens pharmacy within past 12 months)
5. Patient is currently prescribed 5 or more Rx medications (excluding antibiotics); that includes at least one medication from any of the following six therapeutic classes of medications: hyperlipidemia, hypertension, diabetes, multiple sclerosis, hepatitis C, and HIV
6. Patient is primarily responsible for administering own medication

Exclusion Criteria:

1. Severe, uncorrectable vision
2. Hearing impairments
3. Cognitive impairment (as measured by the 6-item screener)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TEAM Strategy: Patients randomized to the TEAM intervention arm will receive at least one call from a Walgreens pharmacist to help them with their complex Rx regimens.TEAM Strategy:
  1. Pharmacists will have read/write EHR access with established Epic security points
  2. Pharmacists will initiate medication reconciliation activities by calling the patient for a Comprehensive Medication Review. Pharmacists will add notes in their medication list for the prescriber, requesting the removal or discontinuation of prescribed drugs that patients report they are not taking and adding medications omitted from the provider's list. The pharmacist will provide notifications via secured Epic messaging direct to prescribers of any patient concerns.
  3. At 6 month if poor adherence is determined, the pharmacist will initiate Therapy Management Review which is a call from the pharmacist to the patient specifically about the medication(s) for which they have poor adherence. If necessary, the pharmacist will create notes and send an in-basket message to the prescriber.
  4. The prescriber will make changes to the patient's EHR and/or contact the patient as they see fit.
Period: Baseline
Arm/Group | TEAM Strategy | Enhanced Usual Care
Started | 61 | 58
Completed | 61 | 58
Not Completed | 0 | 0
Period: 2 Month
Arm/Group | TEAM Strategy | Enhanced Usual Care
Started | 61 | 58
Completed | 54 | 54
Not Completed | 7 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 5 | 3
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: 61 intervention participants initially completed baseline, however one participant was later deemed ineligible and was removed from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | TEAM Strategy | Enhanced Usual Care | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (7.4) | 60.7 (6.3) | 60.8 (60.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 29 | 65
  Male | 24 | 29 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 17 | 34
  White | 40 | 39 | 79
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Interview Language [Count of Participants; unit: Participants]
  English | 28 | 26 | 54
  Spanish | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Medication Reconciliation
Description: Number of medications discrepancies is measured as the sum of omissions (medications listed in the EHR but the patient reported not taking) and commissions (patient reported taking medications not in the EHR) at baseline and 2 months post baseline. Count of discrepancies at the 2 months follow-up is modeled using a multivariate Poisson regression model, with number of prescribed medications as an offset variable. The model is controlled for confounding variables and the number of medication discrepancies at baseline.
  A discrepancy is considered resolved at the 2 month follow-up if the pharmacist indicated the medication to be removed or added to the medication list.
Time Frame: Baseline-2 months
Population: Participants were excluded from the analysis if they were lost to followup at the 2months post baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: number of discrepancies per medication
Groups:
- TEAM Strategy: Patients randomized to the TEAM intervention arm will receive at least one call from a Walgreens pharmacist to help them with their complex Rx regimens.
  TEAM Strategy: 1. Pharmacists will have read/write EHR access with established Epic security points 2. Pharmacists will initiate medication reconciliation activities by calling the patient for a Comprehensive Medication Review. Pharmacists will add notes in their medication list for the prescriber, requesting the removal or discontinuation of prescribed drugs that patients report they are not taking and adding medications omitted from the provider's list. The pharmacist will provide notifications via secured Epic messaging direct to prescribers of any patient concerns.
  3. At 6 month if poor adherence is determined, the pharmacist will initiate Therapy Management Review which is a call from the pharmacist to the patient specifically about the medication(s) for which they have poor adherence. If necessary, the pharmacist will create notes and send an in-basket message to the prescriber.
  4. The prescriber will make changes to the patient's EHR and/or contact the patient as they see fit.
Arm/Group | TEAM Strategy | Enhanced Usual Care
Number analyzed (Participants) | 54 | 54
number of discrepancies per medication | 0.14 [0.08 to 0.23] | 0.17 [0.10 to 0.29]

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | TEAM Strategy | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/58
Other Adverse Events (participants affected / at risk) | 0/61 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT04575155/Prot_SAP_000.pdf